CLINICAL TRIAL: NCT01673334
Title: Prospective Paired Evaluation of EUS-Guided 22 Gauge Core Biopsy Versus Fine-needle Aspiration for Suspected Pancreatic Neoplasms
Brief Title: Evaluation of EUS-Guided 22 Gauge Core Biopsy Versus Fine-needle Aspiration for Suspected Pancreatic Neoplasms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15779
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Tumor
Keywords: Pancreas Tumor EUS FNA Core Biopsy Procore FNB
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fine Needle Aspiration and Core Biospsy (Experimental): Patients will undergo both FNA and core biopsy during EUS evaluation of a solid pancreatic tumor.
  Interventions: Device: Fine Needle Aspiration (FNA) and Core biopsy (FNB)

INTERVENTIONS:
Device: Fine Needle Aspiration (FNA) and Core biopsy (FNB)

SUMMARY:
We aim to compare the efficacy (diagnostic yield), ease of use, and technical success rates of EUS guided 22 gauge fine needle aspiration to core biopsy in the evaluation of pancreatic tumors. The experimental hypothesis is that FNA will have superior overall diagnostic yield than core biopsy.

DETAILED DESCRIPTION:
Background: Endoscopic ultrasonography (EUS) has been utilized for over a decade to evaluate endo-luminal and adjacent tumors of the gastrointestinal tract. In that time, EUS guided fine needle aspiration (FNA) has emerged as the dominant means of tissue acquisition for pancreatic mass lesions. FNA has several limitations, foremost of which is the absence of a clear relationship between cellular elements and stroma which may be required for accurate diagnosis. Additionally, EUS-FNA requires the assistance of an on-site cytopathologist for optimal yield which limits its dissemination and increases its cost. A novel EUS histology needle (EUS-FNB) is available in the 22 gauge diameter which may allow for more accurate diagnosis without the need for on site cytopathology assistance. Aim: To prospectively compare the diagnostic yield, number of needle passes, and ease of use of 22 gauge EUS-FNA and EUS-FNB. Hypothesis: EUS-FNB is superior to traditional EUS-FNA with regard to all primary and secondary outcome measures. Methods: Patients scheduled for EUS evaluation of solid pancreatic tumors will be screened for enrollment at either a preceding clinical encounter or the morning of their scheduled procedure. English-speaking patients between the ages of 18 and 90 with a predominantly solid (greater than 60%) mass lesion of the pancreas will be considered for enrollment. Exclusion criteria include pregnancy, a predominantly cystic lesion, and the presence of an uncorrectable coagulopathy. Patients will then undergo both EUS-FNA and EUS-FNB for the collection of tissue specimens required for clinical care. The results of the experimental approach (EUS-FNB) will be compared to the control approach (EUS-FNA). Data collected for each procedure will include: instrument use order, number of needle passes with each device, technical success of each device, complications, ease of use, and the ultimate pathological diagnosis / diagnostic yield for each device. Each data category will then be compared utilizing standard statistical tests including chi-squared, Fishers' exact, or student's t test.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 90 years.
* Presence of a solid (greater than 60%) mass lesion within the pancreas on cross-sectional imaging, without a preceding tissue diagnosis.
* Absence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not correct with the administration of fresh frozen plasma.
* The patient must read and speak english and has signed informed consent document.
* The patient is scheduled for diagnostic endosonography by their referring provider or UVa gastroenterologist.

Exclusion Criteria:

* Age less than 18 or greater than 90 years.
* The patient is unable to read or understand the consent form.
* The patient is currently pregnant.
* The patient has an uncorrectable coagulopathy as defined by a prolonged prothrombin time (PT) or partial thromboplastin time (PTT) which does not improve with administration of fresh frozen plasma.
* The patient has a pancreatic mass lesion which is predominantly cystic (greater than 40%).
* No mass lesion is identified at the time of endosonography.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-07-09 (Actual); Study Completion 2013-07-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | One-week post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Shami, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States